CLINICAL TRIAL: NCT03546400
Title: A Phase 4, Open-label, Safety, Tolerability And Pharmacokinetic Study Of Methylphenidate Hydrochloride (Hcl) Extended Release Chewable Tablet (Erct) In 4-5 Year Old Children With Attention Deficit Hyperactivity Disorder (Adhd)
Brief Title: Safety, Tolerability and PK Study of Methylphenidate HCl ERCT in 4-5 Year Old Children With ADHD.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was cancelled prior to the enrollment of any participants.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B7491020
Record Dates: First submitted 2018-05-04; First posted 2018-06-06 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- methylphenidate HCl ERCT (Other): methylphenidate HCl ERCT
  Interventions: Drug: methylphenidate HCl ERCT

INTERVENTIONS:
Drug: methylphenidate HCl ERCT — methylphenidate HCl ERCT

SUMMARY:
2-week open-label safety, tolerability and pharmacokinetic study of methylphenidate HCl ERCT in 4-5 year old children with ADHD.

DETAILED DESCRIPTION:
Phase 4, Open-label, Safety, Tolerability And Pharmacokinetic Study Of methylphenidate Hydrochloride (HCl) Extended Release Chewable Tablets (ERCT) In 4-5 Year Old Children With Attention Deficit Hyperactivity Disorder (ADHD)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female child 4-5 years of age at screening.
2. Signed and dated informed consent provided by the subject's parent/legal and assent of the child (as applicable)
3. Meets DSM-5 criteria for ADHD based on the K-SADS-PL.
4. ADHD RS-IV Preschool-Home Version score at Screening and Baseline >/= 90th percentile for gender and age in >/=1 of the following: hyperactive-impulsive subscale, inattentive subscale, or total score.
5. Peabody Picture Vocabulary Test 4 (PPVT-4)Standard Score >/=70.
6. Child Global Assessment Scale (CGAS) score </= 55.
7. History of an adequate course of non medication treatment for ADHD based on investigator judgment or, where such treatments are not available, the severity of the subject's ADHD symptoms are such that medication treatment is deemed necessary by the investigator.

Exclusion Criteria:

1. Treated with atomoxetine within 30 days prior to the Baseline.
2. Received any investigational products or devices within 30 days prior to the Baseline visit.
3. History of stimulant nonresponse, intolerability or hypersensitivity to any dose of methylphenidate or other stimulant.If a subject has a known allergy to D&C red #30, he/she should not be enrolled in the study.
4. An intelligence quotient (IQ) <70.
5. History of acute or chronic medical or psychiatric condition or cardiac or laboratory abnormality.
6. Less than 5th percentile for height or weight at Screening.
7. History of recent clinically significant self-harming behaviors.

Ages: 48 Months to 69 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-09-25 (Estimated); Primary Completion 2020-12-03 (Estimated); Study Completion 2020-12-03 (Estimated)

PRIMARY OUTCOMES:
PK parameter-Tmax | 2 weeks
  PK profile of methylphenidate following a single oral dose of 30 mg methylphenidate HCl ERCT.
PK parameter- Cmax | 2 weeks
  PK profile of methylphenidate following a single oral dose of 30 mg methylphenidate HCl ERCT.
PK parameter- AUClast | 2 weeks
  PK profile of methylphenidate following a single oral dose of 30 mg methylphenidate HCl ERCT.
PK parameter-AUC0-2 | 2 weeks
  PK profile of methylphenidate following a single oral dose of 30 mg methylphenidate HCl ERCT.
PK parameter-AUC2-6 | 2 weeks
  PK profile of methylphenidate following a single oral dose of 30 mg methylphenidate HCl ERCT.
PK parameter-AUC6-24 | 2 weeks
  PK profile of methylphenidate following a single oral dose of 30 mg methylphenidate HCl ERCT.
PK parameter-AUCinf | 2 weeks
  PK profile of methylphenidate following a single oral dose of 30 mg methylphenidate HCl ERCT.
PK parameter- t1/2 | 2 weeks
  PK profile of methylphenidate following a single oral dose of 30 mg methylphenidate HCl ERCT.
PK parameter-CL/F | 2 weeks
  PK profile of methylphenidate following a single oral dose of 30 mg methylphenidate HCl ERCT.
PK parameter-Vz/F | 2 weeks
  PK profile of methylphenidate following a single oral dose of 30 mg methylphenidate HCl ERCT.

SECONDARY OUTCOMES:
incidence of treatment emergent adverse events (safety and tolerability) | 2 weeks
  incidence of treatment emergent adverse events (safety and tolerability)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7491020&StudyName=An+Open+Label+Pharmacokinetic+Study+Of+Methylphenidate+Extended+Release+Chewable+Tablet+%28erct%29+In+Adhd+Patients+Aged+4-5+Years+Old
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7491020&StudyName=A+Phase+4%2C+Open+Label%2C+Safety%2C+Tolerability+And+Pharmacokinetic+Study+Of+Quillichew+Extended+Release+Chewable+Tablets+%28methylphenidate+Hcl+Extended+Release+Chewable+Tablets+%5Berct%5D%29+In+4+5+Year+Old+Children+With+Attention+Deficit+Hyperactivity+Disorder+%28adhd%29
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7491020&StudyName=A+Phase+4%2C+Open-label%2C+Safety%2C+Tolerability+And+Pharmacokinetic+Study+Of+Quillichew+%28methylphenidate+Hydrochloride+%28hcl%29%29+Extended+Release+Chewable+Tablets+%28erct%29+In+4+5+Year+Old+Children+With+Attention+Deficit+Hyperactivity+Disorder+%28adhd%29
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7491017&StudyName=A+Multi-center%2C+Double-blind%2C+Randomized%2C+Placebo-controlled%2C+Parallel+Group+Study+Evaluating+The+Safety+And+Efficacy+Of+Quillivant+Xr+In+The+Treatment+Of+Pre-school+Aged+Children+With+Adhd
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7491017&StudyName=A+Phase+4%2C+Double-blind%2C+Randomized%2C+Parallel+Group%2C+Placebo-controlled+Study+Of+The+Efficacy+And+Safety+Of+Quillichew+Extended+Release+Chewable+Tablets+%28methylphenidate+Hcl+Extended+Release+Chewable+Tablets+%28erct%29%29++In+4-5+Year+Old+Children+With+Attention+Deficit+Hyperactivity+Disorder+%28adhd%29.
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7491017&StudyName=A+Phase+4%2C+Double-blind%2C+Randomized%2C+Parallel+Group%2C+Placebo-controlled+Study+Of+The+Efficacy+And+Safety+Of+Quillichew+%28methylphenidate+Hydrochloride+%28hcl%29%29+Extended+Release+Chewable+Tablets+%28erct%29+In+4-5+Year+Old+Children+With+Attention+Deficit+Hyperactivity+Disorder+%28adhd%29
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7491020&StudyName=A+Phase+4%2C+Open-label%2C+Safety%2C+Tolerability+And+Pharmacokinetic+Study+Of+Methylphenidate+Hydrochloride+%28hcl%29+Extended+Release+Chewable+Tablet+%28erct%29+In+4-5+Year+Old+Children+With+Attention+Deficit+Hyperactivity+Disorder+%28adhd%29